CLINICAL TRIAL: NCT02254369
Title: A Randomized, Phase 1, Double-Blind, Placebo-Controlled, First-in-Human, Safety, Tolerability, and Pharmacokinetic Study of Single Ascending Doses of GC021109 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of Single Ascending Doses of GC021109 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GliaCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC-100-01
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (10):
- Cohort 1- GC021109 (Experimental): single dose, 0.0014 mg/kg GC021109
  Interventions: Drug: GC021109
- Cohort 2- GC021109 (Experimental): single dose, 0.014 mg/kg GC021109
  Interventions: Drug: GC021109
- Cohort 3-GC021109 (Experimental): single dose, 0.14 mg/kg GC021109
  Interventions: Drug: GC021109
- Cohort 4- GC021109 (Experimental): single dose, 1.4 mg/kg GC021109 subjects will receive GC021109 under fasting then under fed conditions separated by a washout of 14 (± 1) days after the first dose.
  Interventions: Drug: GC021109
- Cohort 5- GC021109 (Experimental): single dose, 4.2 mg/kg GC021109
  Interventions: Drug: GC021109
- Cohort 1- placebo (Placebo Comparator): single dose, 0.0014 mg/kg matching placebo
  Interventions: Other: Placebo
- Cohort 2- placebo (Placebo Comparator): single dose, 0.014 mg/kg matching placebo
  Interventions: Other: Placebo
- Cohort 3- placebo (Placebo Comparator): single dose, 0.14 mg/kg matching placebo
  Interventions: Other: Placebo
- Cohort 4- placebo (Placebo Comparator): single dose, 1.4 mg/kg subjects will receive matching placebo under fasting then under fed conditions separated by a washout of 14 (+/- 1) days after the first dose.
  Interventions: Other: Placebo
- Cohort 5- placebo (Placebo Comparator): single dose, 4.2 mg/kg matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GC021109
  Arms: Cohort 1- GC021109; Cohort 2- GC021109; Cohort 3-GC021109; Cohort 4- GC021109; Cohort 5- GC021109
Other: Placebo
  Arms: Cohort 1- placebo; Cohort 2- placebo; Cohort 3- placebo; Cohort 4- placebo; Cohort 5- placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of single oral doses of GC021109 when administered to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or non-childbearing potential females, 18 to 55 years of age, inclusive, at the time of informed consent.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to dosing of study drug.
3. BMI ≥ 18.5 and ≤ 32.0 (kg/m2) at screening with a maximum weight of 120 kg.
4. Medically healthy with no clinically significant screening results that would exclude subject from the study as deemed by the PI.
5. Females must have undergone 1 of the following sterilization procedures, and have official documentation, at least 6 months prior to dosing of study drug:

   * Hysteroscopic sterilization
   * Bilateral tubal ligation or bilateral salpingectomy
   * Hysterectomy.
   * Bilateral oophorectomy. OR be postmenopausal with amenorrhea for at least 1 year prior to dosing of study drug and have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
6. All male subjects must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug.
7. If male, must agree to not donate sperm from Day -1 until 90 days after dosing.
8. Understand the study procedures in the ICF, and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History of any illness that, in the opinion of the PI, might confound the results of the study or pose an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to screening.
5. History or presence of hypersensitivity or idiosyncratic reaction to component of the study drug or related compounds.
6. History of cancer within the past 5 years (excluding non-melanoma skin cancer) prior to screening.
7. Clinically significant abnormal screening laboratory test values (as determined by the

   PI), including, but not limited to, the following:
   * any values for alanine aminotransferase (ALT) or aspartate aminotransferase (AST) that are above the upper limit of the reference range at screening or check-in.
   * any values for total or direct bilirubin that are 1.5 times above the upper limit of the reference range at screening or check-in.
   * estimated creatinine clearance <90 mL/min at screening only.
8. Clinically significant infection within 3 months prior to screening as determined by the PI.
9. Female subjects of child-bearing potential.
10. Female subjects who are pregnant or lactating.
11. Positive urine drug or urine alcohol results at screening or check-in.
12. Positive urine cotinine at screening.
13. Positive results at screening for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
14. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
15. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
16. Orthostatic vital sign results as deemed clinically significant in the opinion of the PI at screening.
17. QTcB interval is >430 msec (males) or >450 msec (females) or deemed clinically abnormal by the PI, prior to dosing of study drug.
18. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non-prescription medications, herbal remedies, vitamin supplements or substrates of CYP1A2, CYP3B6, or CYP3A4 beginning 14 days prior to dosing of study drug and throughout the study. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study.
    * Any drugs known to be significant inducers of CYP enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, for 28 days prior to dosing of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/PD interaction with study drug.
19. Has been on a diet incompatible with the on-study diet, in the opinion of the PI, within the 28 days prior to dosing of study drug, and throughout the study.
20. Has donated blood within 3 months of screening visit or plans to donate blood within 3 months of study completion, except for blood collected during another clinical trial performed 30 days prior to screening.
21. Plasma donation within 7 days prior to dosing of study drug.
22. Participation in another clinical trial within 30 days prior to screening. The 30-day window will be derived from the date of the last study scheduled blood collection or dosing, whichever is later, in the previous study to the date of screening for the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number and severity of TEAEs | following single dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Neptune City, New Jersey, United States